CLINICAL TRIAL: NCT01910675
Title: Use of Prothrombin Complex Concentrate and Fibrinogen Compared With Fresh Frozen Plasma (and Fibrinogen if Needed) in the Treatment of Postpartum Haemorrhage
Brief Title: PCC and Fibrinogen Compared With FFP in PPH
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Impossible to get a written informed consent beforehand
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jouni Ahonen, Consultant anaesthesiologist, M.D., Ph.D., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT-2012-003128; U1030N7560 (Other: HUCH)
Record Dates: First submitted 2013-07-13; First posted 2013-07-30 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Postpartum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — prothrombin complex concentrates

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PCC group (Experimental): Twenty patients in the PCC group receive 15 IU/kg of Octaplex concentrate and 2 g of Riastap concentrate. Additional fibrinogen is administered (if needed) to increase the baseline FIBTEM-MCF (at 5 min) to the target of 15 mm.
  Interventions: Drug: PCC
- FFP group (Active Comparator): Twenty patients in the FFP group receive 4 units of FFP (Octaplas). Additional fibrinogen (Riastab) is administered (if needed) to increase the baseline FIBTEM-MCF (at 5 min) to the target of 15 mm. The fibrinogen content of the FFP will be taken into consideration (2.1 g in 4 units of FFP).
  Interventions: Drug: FFP

INTERVENTIONS:
Drug: PCC — 15 IU/kg Octaplex and 2 g Riastab. Additional fibrinogen if needed.
  Other Names: Octaplex, Riastab
  Arms: PCC group
Drug: FFP — 4 units Octaplas. Additional fibrinogen if needed.
  Other Names: Octaplas
  Arms: FFP group

SUMMARY:
The purpose of the study is to find out if the regimen of prothrombin complex concentrate (PCC) together with fibrinogen concentrate is as efficient as fresh frozen plasma (FFP) (plus fibrinogen if needed) during the early stages of the transfusion therapy in postpartum haemorrhage (PPH). The original protocol included the use of HES and the recruitment of patients was postponed while waiting the final decision by EMA. All HES solutions were abandoned at our institution in September and an amendment was made to change the protocol. HES solution are replaced by the use of hyperoncotic (20%) albumin.

DETAILED DESCRIPTION:
Forty patients are randomized to receive either PCC and fibrinogen concentrate (PCC group) or FFP (and fibrinogen if needed) (FFP group), 20 patients in each group. Patients in the PCC group receive 15 IU/kg of PCC concentrate and 2 g of fibrinogen concentrate. Patients in the FFP group receive 4 units of FFP. In both groups, additional fibrinogen is administered (if needed) to increase the baseline FIBTEM-MCF (at 5 min) to the target of 15 mm.

Baseline blood samples will be drawn at study inclusion when the (on-going) blood loss exceeds 1500 ml. The next samples will be drawn at 45 min (or immediately after the administration of the study drug if later). Otherwise, the management protocol strictly follows the local PPH guideline.

The primary endpoint is the amount of blood loss within the first 6 and 24 hours after delivery. Secondary endpoints include the difference/similarity in the laboratory determinations (ia coagulation screen, PFA-100, CAT and ROTEM).

ELIGIBILITY:
Inclusion Criteria:

Women who have delivered vaginally or by caesarean section with a PPH of 2000 ml (the amount of blood loss: in addition to the suctioned blood, sponges, wraps, swabs, etc. are carefully weighed)

Exclusion Criteria:

Women with a history of bleeding tendency or hepatic or renal insufficiency, or PPH exceeding 3000 ml because in that case the initial need for fibrinogen may be even more

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Blood loss | Within the first 6 and 24 hours after delivery
  The suctioned blood is recorded and sponges, wraps, swabs, etc. are carefully weighed. The amount of blood loss will be compared between the groups.

SECONDARY OUTCOMES:
Maximum clot firmness (MCF) | At the time when the blood loss exceeds 1500 ml and 45 min later
  INTEM, EXTEM, FIBTEM and APTEM / ROTEM
Endogenous thrombin potential | At the time when the blood loss exceeds 1500 ml and 45 min later
  CAT
Fibrinogen level | At the time when the blood loss exceeds 1500 ml and 45 min later
  Clauss method
Platelet function | At the time when the blood loss exceeds 1500 ml and 45 min later
  PFA-100
Clotting time (CT) | At the time when the blood loss exceeds 1500 ml and 45 min later
  INTEM, EXTEM, FIBTEM and APTEM / ROTEM
Clot formation time (CFT) | At the time when the blood loss exceeds 1500 ml and 45 min later
  INTEM, EXTEM, FIBTEM and APTEM / ROTEM

CONTACTS AND LOCATIONS:
Overall Officials: Jouni V. Ahonen, Ph.D., M.D., Principal Investigator — Maternity Hospital, Helsinki University Central Hospital
Locations (1):
- Maternity Hospital, Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

REFERENCES:
- [Background] Ahonen J, Stefanovic V, Lassila R. Management of post-partum haemorrhage. Acta Anaesthesiol Scand. 2010 Nov;54(10):1164-78. doi: 10.1111/j.1399-6576.2010.02309.x. PMID 21069897